CLINICAL TRIAL: NCT02943954
Title: FLOW Evaluation to Guide Revascularization in Multi-vessel ST-elevation Myocardial Infarction
Acronym: FLOWER-MI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Abbott (Industry); Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P150943; 2016-A00418-43 (Other: Agence Nationale de Securite du Medicament et des Produits de Sante); AOM15608 (Other Grant/Funding Number: French Ministry of Health)
Record Dates: First submitted 2016-09-07; First posted 2016-10-25 (Estimated); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Acute ST Segment Elevation Myocardial Infarction; Acute Myocardial Infarction; Multi Vessel Coronary Artery Disease
Keywords: Fractional Flow Reserve
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Angiography guided PCI (Other): Revascularisation of non-culprit lesions guided by PCI
  Interventions: Procedure: Angiography guided PCI
- FFR guided PCI (Other): Revascularisation of non-culprit lesions guided by FFR measurement
  Interventions: Device: Fractional Flow Reserve (FFR)

INTERVENTIONS:
Procedure: Angiography guided PCI
  Arms: Angiography guided PCI
Device: Fractional Flow Reserve (FFR)
  Arms: FFR guided PCI

SUMMARY:
Although current guidelines recommend fractional flow reserve (FFR) to identify haemodynamically relevant coronary lesion(s) in stable patients when evidence of ischaemia is not available (Class I, Level of Evidence: A), no published study has assessed the usefulness of FFR to guide percutaneous coronary intervention (PCI) in ST-elevation myocardial infarction (STEMI) patients with multi-vessel disease (MVD).

The main objective of this study is to determine whether, in STEMI patients with MVD amenable to PCI, the use of FFR in addition to angiography will improve cardiovascular outcomes, compared with the current practice of angiography- guided PCI, by improving the appropriateness of revascularisations by assessing the relevance of non-culprit lesions in the context of STEMI with multivessel coronary artery disease.

The secondary objective is to assess the safety and the cost-effectiveness of the FFR-guided strategy compared to the angiography-guided strategy.

DETAILED DESCRIPTION:
The optimal revascularisation strategy in STEMI patients with MVD is currently debated. Recent data suggest that MV-PCI may be the most appropriate option for treating such patients. Consequently, the real challenge becomes to define what MVD is, in the context of acute MI, in order to limit revascularisation by PCI to vessels that truly need it. Visual estimation of the degree of coronary stenoses is a poor indicator of their haemodynamic severity. FFR is precisely designed and recommended in current guidelines to provide objective guidance for the functional assessment of lesion severity during coronary angiography in stable patients, but it has not been validated in STEMI patients with MVD. The purpose of the present trial will therefore be to investigate the relevance of FFR to guide the revascularisation management of patients at the acute stage of STEMI.

STEMI patients with successful culprit lesion PCI (primary, rescue or pharmaco-invasive) and ≥ 50% diameter stenosis by visual estimate, in which revascularization is contemplated and judged amenable to PCI in at least one additional non-culprit lesion will be randomized into two groups: angiography-guided PCI or FFR-guided PCI.

If the patient is randomized to the angiography-guided PCI, all the lesions indicated beforehand will be treated. If the patient is randomized to the FFR-guided PCI, measurements of FFR of non-infarct related lesion(s) will be performed and only those lesions with a FFR ≤ 0.80 will be treated.

The use of drug-eluting stents is encouraged in both strategies. All patients will receive optimal medical therapy (including dual antiplatelet therapy, beta-blockers, statins, ACE-I or ARB) as recommended in international guidelines in both strategies.

Clinical follow-up will be performed at discharge, 30-day, 6 month and one-year. Rates of major adverse cardiac events, functional class and number of anti-anginal medications used will be collected. If the patient has been rehospitalized since index hospital discharge, the discharge summary and all relevant information will be collected.

ELIGIBILITY:
Inclusion Criteria:

* STEMI patients ≥ 18 years old with successful culprit lesion PCI (primary, rescue or pharmaco-invasive) and ≥ 50% stenosis judged amenable to PCI in at least one additional non-culprit lesion
* Written informed consent

Exclusion Criteria:

* Patients with cardiogenic shock (SBP < 90 mmHg with clinical signs of low output or patients requiring inotropic agents)
* Patients with MVD referred to surgery for CABG or treatment of acute complications (e.g. ventricular septal rupture)
* Patients with one-vessel disease
* Previous coronary bypass surgery
* Extremely tortuous, calcified coronary vessels or chronic total occlusion (CTO)
* Life expectancy < 2 years
* Patients with known hypersensitivity to adenosine
* Pregnancy
* Participation in another interventional therapeutic study at the same time or within 3 months prior to the beginning of the present study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1170 (Estimated)
Dates: Start 2016-12 (Actual); Primary Completion 2020-10-24 (Actual); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Rate of major adverse cardiac events | 1 year
  Number of deaths, myocardial infarctions and unplanned hospitalization leading to urgent revascularizations at one year.

SECONDARY OUTCOMES:
Deaths | 1 year
Myocardial infarctions | 1 year
Repeat revascularizations | 1 year
Rate of nonculprit artery target lesion treated by urgent revascularization | 1 year
Rates of major adverse cardiac events at 30 days and 6 months | 30 days and 6 months
Rehospitalization for angina during the follow up period | 1 year
Procedure time | 5 days
Functional class at 1 year | 1 year
  The functional class is assessed with the use of the Canadian Cardiovascular Society classification of angina.
Health-related quality of life | 1 year
  Health-related quality of life is assessed by the European Quality of Life-5 Dimensions [EQ-5D] questionnaires
Anti-anginal medications used | 1 month, 6 months and 1 year
  Number of anti-anginal medications used
Cost effectiveness | 1 year
  Incremental cost effectiveness ratio (ICER) using the composite endpoint (all-cause death, myocardial infarctions and repeat revascularizations).
Cost utility | 1 year
  Incremental cost-utility ration (ICUR) using quality-adjusted life years (QALYs)

CONTACTS AND LOCATIONS:
Overall Officials: Etienne PUYMIRAT, MD, Principal Investigator — AP - HP, Hôpital Europeen Georges-Pompidou, Paris, France
Locations (1):
- France, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Authors/Task Force members; Windecker S, Kolh P, Alfonso F, Collet JP, Cremer J, Falk V, Filippatos G, Hamm C, Head SJ, Juni P, Kappetein AP, Kastrati A, Knuuti J, Landmesser U, Laufer G, Neumann FJ, Richter DJ, Schauerte P, Sousa Uva M, Stefanini GG, Taggart DP, Torracca L, Valgimigli M, Wijns W, Witkowski A. 2014 ESC/EACTS Guidelines on myocardial revascularization: The Task Force on Myocardial Revascularization of the European Society of Cardiology (ESC) and the European Association for Cardio-Thoracic Surgery (EACTS)Developed with the special contribution of the European Association of Percutaneous Cardiovascular Interventions (EAPCI). Eur Heart J. 2014 Oct 1;35(37):2541-619. doi: 10.1093/eurheartj/ehu278. Epub 2014 Aug 29. No abstract available. PMID 25173339
- [Background] Tonino PA, De Bruyne B, Pijls NH, Siebert U, Ikeno F, van' t Veer M, Klauss V, Manoharan G, Engstrom T, Oldroyd KG, Ver Lee PN, MacCarthy PA, Fearon WF; FAME Study Investigators. Fractional flow reserve versus angiography for guiding percutaneous coronary intervention. N Engl J Med. 2009 Jan 15;360(3):213-24. doi: 10.1056/NEJMoa0807611. PMID 19144937
- [Background] Ntalianis A, Sels JW, Davidavicius G, Tanaka N, Muller O, Trana C, Barbato E, Hamilos M, Mangiacapra F, Heyndrickx GR, Wijns W, Pijls NH, De Bruyne B. Fractional flow reserve for the assessment of nonculprit coronary artery stenoses in patients with acute myocardial infarction. JACC Cardiovasc Interv. 2010 Dec;3(12):1274-81. doi: 10.1016/j.jcin.2010.08.025. PMID 21232721
- [Background] Engstrom T, Kelbaek H, Helqvist S, Hofsten DE, Klovgaard L, Holmvang L, Jorgensen E, Pedersen F, Saunamaki K, Clemmensen P, De Backer O, Ravkilde J, Tilsted HH, Villadsen AB, Aaroe J, Jensen SE, Raungaard B, Kober L; DANAMI-3-PRIMULTI Investigators. Complete revascularisation versus treatment of the culprit lesion only in patients with ST-segment elevation myocardial infarction and multivessel disease (DANAMI-3-PRIMULTI): an open-label, randomised controlled trial. Lancet. 2015 Aug 15;386(9994):665-71. doi: 10.1016/s0140-6736(15)60648-1. PMID 26347918
- [Derived] Puymirat E, Cayla G, Simon T, Steg PG, Montalescot G, Durand-Zaleski I, Ngaleu Siaha F, Gallet R, Khalife K, Morelle JF, Motreff P, Lemesle G, Dillinger JG, Lhermusier T, Silvain J, Roule V, Labeque JN, Range G, Ducrocq G, Cottin Y, Blanchard D, Charles Nelson A, Djadi-Prat J, Chatellier G, Danchin N; FLOWER-MI Study Investigators. Three-Year Outcomes With Fractional Flow Reserve-Guided or Angiography-Guided Multivessel Percutaneous Coronary Intervention for Myocardial Infarction. Circ Cardiovasc Interv. 2024 Jun;17(6):e013913. doi: 10.1161/CIRCINTERVENTIONS.123.013913. Epub 2024 May 24. PMID 38785084
- [Derived] Denormandie P, Simon T, Cayla G, Steg PG, Montalescot G, Durand-Zaleski I, le Bras A, le Breton H, Valy Y, Schiele F, Cuisset T, Vanzetto G, Levesque S, Goube P, Nallet O, Angoulvant D, Roubille F, Charles Nelson A, Chatellier G, Danchin N, Puymirat E. Compared Outcomes of ST-Segment-Elevation Myocardial Infarction Patients With Multivessel Disease Treated With Primary Percutaneous Coronary Intervention and Preserved Fractional Flow Reserve of Nonculprit Lesions Treated Conservatively and of Those With Low Fractional Flow Reserve Managed Invasively: Insights From the FLOWER-MI Trial. Circ Cardiovasc Interv. 2021 Nov;14(11):e011314. doi: 10.1161/CIRCINTERVENTIONS.121.011314. Epub 2021 Aug 23. PMID 34420366
- [Derived] Puymirat E, Cayla G, Simon T, Steg PG, Montalescot G, Durand-Zaleski I, le Bras A, Gallet R, Khalife K, Morelle JF, Motreff P, Lemesle G, Dillinger JG, Lhermusier T, Silvain J, Roule V, Labeque JN, Range G, Ducrocq G, Cottin Y, Blanchard D, Charles Nelson A, De Bruyne B, Chatellier G, Danchin N; FLOWER-MI Study Investigators. Multivessel PCI Guided by FFR or Angiography for Myocardial Infarction. N Engl J Med. 2021 Jul 22;385(4):297-308. doi: 10.1056/NEJMoa2104650. Epub 2021 May 16. PMID 33999545
- [Derived] Puymirat E, Simon T, de Bruyne B, Montalescot G, Steg G, Cayla G, Durand-Zaleski I, Blanchard D, Danchin N, Chatellier G; FLOWER-MI study investigators. Rationale and design of the Flow Evaluation to Guide Revascularization in Multivessel ST-Elevation Myocardial Infarction (FLOWER-MI) trial. Am Heart J. 2020 Apr;222:1-7. doi: 10.1016/j.ahj.2019.12.015. Epub 2019 Dec 27. PMID 32000067